CLINICAL TRIAL: NCT03287752
Title: A Prospective Randomized Comparison of the Effect of BASKA Mask Versus Endo Tracheal Tube on Respiratory Function Parameters in Patients Undergoing Gynecological Laparoscopic Surgery
Brief Title: BASKA Mask Versus Endo Tracheal Tube in Gynecological Laparoscopic Surgery
Acronym: BASKAMASK
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Other Study IDs: 17100178
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BASKA MASK: Patients will be anesthetized using BASKA mask after lubrication with water soluble lubricant.
  Interventions: Device: BASKA MASK
- Endotracheal tube: Patients will be anesthetized using appropriate sized cuffed oral endotracheal tube ETT.
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: BASKA MASK — Patients will be anesthetized using BASKA mask after lubrication with water soluble lubricant
  Other Names: BASKA
  Groups: BASKA MASK
Device: Endotracheal tube — Patients will be anesthetized using appropriate sized cuffed oral endotracheal tube.
  Other Names: ETT
  Groups: Endotracheal tube

SUMMARY:
The BASKA mask (Logikal Health Products PTY Ltd., Morisset, NSW, Australia) is a novel supraglottic airway device. It has many of the features of other supraglottic airways, with a number of innovations. These include; A non-inflatable cuff, that it is continuous with the central channel of the device. As the pressure increases with positive pressure ventilation, the cuff itself is 'inflated', this may improve the seal, reduce leak, and make ventilation more efficient.

DETAILED DESCRIPTION:
The BASKA mask incorporates an inlet that fits into the upper esophagus, and the dorsal surface of the cuff is moulded to direct any oropharyngeal contents away from the glottis and towards the side channels to which suction can be attached to facilitate aspiration of this space (Fig.1c). These features may reduce the risk of pulmonary aspiration of secretions or gastric contents that accumulate in the supraglottic area.

Compared with previous versions, these modifications have made BASKA mask airway a fairly safe and effective airway device in low-risk patients undergoing gynecologic laparoscopic surgeries

ELIGIBILITY:
Inclusion Criteria:

Sex: Female patients scheduled for elective gynecological laparoscopic surgery.

* Age: 18-60 years.
* BMI< 30kg/m2.
* ASA physical status: I-II.
* Operation: gynecological laparoscopic surgery under general anesthesia of an anticipated duration<1h.

Exclusion Criteria:

* Patient refusal.
* History of cardiac disease, psychological disorders, respiratory diseases including asthma, renal or hepatic failure.
* Patients who have high risk of regurgitation or aspiration based on history of gastro esophageal reflux, hiatus hernia, diabetes and gross obesity.
* Neck pathology.
* Patients who predicted difficult airway (based on a history of difficult airway, mouth opening was less than 2.5 cm, inter-incisor distance < 20 mm, cervical spine pathology, modified Mallampati class III/IV, or thyromental distance < 65 mm).
* Allergy to any of the anesthetic agents used.
* The possibility of being pregnant.
* Heavy smoker.
* Preoperative sore throat.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females 18-60years
Study Population: Female patients scheduled for elective gynecological laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
Peak airway pressure | 6 hours including preoperative, intraoperative and 4h after operation
  Peak airway pressure before and after abdominal inflation.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Assisstant professor in anesthesia and intensive care, faculty of medicine, Assiut university, Egypt
Locations (1):
- women health hospital, Assiut university, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No